CLINICAL TRIAL: NCT06216522
Title: A Randomised-controlled Trial on the Effectiveness of Topical Sesame Oil in Preventing Phlebitis at Intravenous Cannula Sites in Adult Patients
Brief Title: The Effectiveness of Topical Sesame Oil in Preventing Phlebitis at IV Cannula Sites in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021/2804
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Phlebitis; Thrombophlebitis
Keywords: intravenous cannula; IV cannula; Adult; Cardiovascular; Cardiothoracic; Phlebitis; Thrombophlebitis
MeSH Terms: conditions — Phlebitis; Thrombophlebitis | interventions — Sesame Oil; Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 5 drops/0.25mls of 100% sesame oil will be applied to the IV cannula site, from 3cm above the insertion point to 10cm along the vein, with a width of 2cm on either side, every 12 hours for 72 hours.
  Interventions: Other: Topical Sesame Oil
- Control (Placebo Comparator): 5 drops/0.25mls of liquid paraffin oil will be applied to the IV cannula site, from 3cm above the insertion point to 10cm along the vein, with a width of 2cm on either side, every 12 hours for 72 hours.
  Interventions: Other: Liquid paraffin oil

INTERVENTIONS:
Other: Topical Sesame Oil — 5 drops/0.25mls of sesame oil applied to the IV cannula site at 12 hourly intervals for 72 hours
  Arms: Intervention
Other: Liquid paraffin oil — 5 drops/0.25mls of liquid paraffin oil applied to the IV cannula site at 12 hourly intervals for 72 hours
  Arms: Control

SUMMARY:
The goal of this randomised controlled trial is to determine the effectiveness of topical sesame oil in preventing phlebitis at peripheral intravenous (IV) cannula sites in adult patients within a cardiovascular and cardiothoracic department of a tertiary hospital.

The main question it aims to answer is:

Is topical sesame oil effective in preventing phlebitis at peripheral IV cannula sites in adult patients within a cardiovascular and cardiothoracic department of a tertiary hospital?

Participants will be randomly allocated to the experimental or control group with the use of a randomisation software (MS excel). They will each have five drops/0.25mls of 100% sesame oil (experimental) or liquid paraffin oil (control) applied to the IV cannula site, at 12 hourly intervals for a total of 72 hours, from 3cm above the insertion point to 10cm along the vein, with a width of 2cm on either side.

Researchers will compare the phlebitis incidence and severity of each group to see if topical sesame oil is more effective than liquid paraffin oil in preventing phlebitis at IV cannula sites in adult patients within a cardiovascular and cardiothoracic department of a tertiary hospital.

DETAILED DESCRIPTION:
The goal of this randomised controlled trial is to determine the effectiveness of topical sesame oil in preventing phlebitis at peripheral intravenous (IV) cannula sites in adult patients within a cardiovascular and cardiothoracic department of a tertiary hospital.

All newly admitted patients with an existing IV cannula will be approached after being admitted into an inpatient ward. This will take place within 12 hours of the IV cannula insertion. They will not be approached if in distress, drowsy or immediately prior to a surgical procedure. The IV cannula will be tested for patency, and assessed for redness, swelling, pain, a palpable venous cord or pyrexia. If any of these symptoms are present, or if the IV cannula is not patent, the recruitment will be terminated.

Participants will be randomly allocated to the experimental or control group with the use of a randomisation software (MS excel). They will each have five drops/0.25mls of 100% sesame oil (experimental) or liquid paraffin oil (control) applied to the IV cannula site, at 12 hourly intervals for a total of 72 hours, from 3cm above the insertion point to 10cm along the vein, with a width of 2cm on either side.

Demographic and clinical data will be recorded into a table. The patient will be instructed not to wash or wipe the topical agent off. The time and date of the start of treatment applied and subsequent treatments at 12 hour intervals will be documented. At the start of the study and at each 12 hour interval, the investigator will observe for signs of phlebitis using the modified Visual Infusion Phlebitis (VIP) scoring tool (1), before application of the next treatment. The study investigators will be the only ones applying the treatment/control and completing the data collection form every 12 hours.

Application of the treatment or control will be made every 12 hours for up to 72 hours, where the IV cannula will then be removed according to hospital guidelines. The IV cannula site will be observed, every 12 hours for up to 24 hours post IV cannula removal, for phlebitis or complications.

Patients will be withdrawn from the study the moment they show signs of adverse reactions from the topical treatment or control.

Participants will be involved in the study for a maximum of 96 hours. If the IV cannula is removed accidentally or not due to phlebitis before the 72-hour period is up, re-insertion of a new cannula and re-application of oils will not be done on a new site.

The application of either sesame oil or liquid paraffin oil is not part of the routine procedures or standard of care in the ward, and will only be applied for the purpose of this research. Both the sesame oil and liquid paraffin oil are marketed products and will be used as per label.

All hardcopy research data will be stored in in a locked cupboard with lock and key access within the National Heart Centre, Singapore. All soft copies will be stored in a password protected Laptop belonging to the principal investigator. Only the principal investigator will have access to the research data. All other members of the research team will access the data through the principal investigator. The physical research data will be kept under lock and key for 7 years after the completion of the research study or date of publication of the research using the research data, whichever is later. After which, all data will be destroyed. Hardcopies will be shredded and soft copies will be deleted.

Subjects may withdraw voluntarily from participation in the study at any time. Subjects may also withdraw voluntarily from receiving the study intervention for any reason. Upon withdrawal, IV cannula sites will continue to be observed for 24 hours at 12-hour intervals for potential reactions to the oils or signs of phlebitis. If there are any adverse reactions to the oils or signs of phlebitis during the 24-hour observation period, the patient will be referred to the attending physician and medical treatment will be rendered. The patient will continue to receive follow-up and medical treatment until symptoms have resolved.

The study may be discontinued at any time, if safety issues arise. If the risks to participants unexpectedly outweigh the benefits due to unexpected severe adverse events due to the application of the treatment or control oils, the study may then be suspended until the risk-benefit ratio is re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80
* Patients must speak and understand either English or Mandarin
* Patients who possess a peripheral IV cannula
* IV cannula must have been inserted for less than 12 hours
* IV cannula must be on an upper extremity
* IV cannula must be patent
* IV cannula sites must show no signs of redness, swelling, pain, a palpable venous cord or pyrexia
* Patient must be admitted to a cardiology ward in the National Heart Centre Singapore

Exclusion Criteria:

* Patients who do not speak or understand either English or Mandarin
* Patients with venous insufficiency
* Patients with coagulopathies
* Patients with cognitive or sensory impairments that would inhibit their ability to rate their pain via a Numerical Rating Scale (NRS)
* Patients who are receiving medications that might interfere with timely reporting of adverse events (eg. medications that cause severe drowsiness)
* Patients who report allergies to sesame or liquid paraffin oil
* IV cannulas that were inserted and used for resuscitation
* Patients with existing skin conditions that cause their skin to be red or swollen and might affect the investigators ability to assess for phlebitis
* Patients who possess more than one peripheral IV cannula will only be included in the study once. All subsequent IV cannula insertions will be excluded.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Phlebitis incidence | At 12 hourly intervals for a total of 72 hours
  Measuring the incidence of phlebitis across both the intervention and control groups

SECONDARY OUTCOMES:
Phlebitis severity | At 12 hourly intervals for a total of 72 hours
  Documenting the severity of phlebitis using the Visual Infusion Phlebitis (VIP) scoring tool, across both the intervention and control groups. It is rated on a scale of zero to five, with five being the worst possible outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Tan, Principal Investigator — Nanyang Polytechnic
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson A. Infection control--a battle in vein: infusion phlebitis. Nurs Times. 1998 Jan 28-Feb 3;94(4):68, 71. No abstract available. PMID 9510815

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT06216522/Prot_SAP_000.pdf